CLINICAL TRIAL: NCT04825444
Title: Clinical Study of Vascular Imaging Evaluation of Computed Tomography Photoacoustic Breast Imaging System
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Union Photoacoustic technologies Co., Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: KND-QX-CXXT
Record Dates: First submitted 2021-03-28; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Breast Tumor; Ultrasonography
Keywords: photoacoustic imaging; Ultrasonography; Breast Tumor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Photoacoustic inspection — Use photoacoustic imaging system to image breast blood vessels

SUMMARY:
Using color Doppler ultrasound to screen people with breast masses. For the patients who show only a single mass on either side of the breast in color Doppler ultrasound, computer tomography photoacoustic breast imaging will be performed. By comparing the two modalities, the blood vessel imaging performance of the computer tomography photoacoustic breast imaging system developed by Union Photoacoustic technologies Co., Ltd is evaluated.

The evaluation index of this experiment is the percentage of blood vessel pixels in the same region of interest (Region Of Interest, ROI) to the total area of the ROI.

DETAILED DESCRIPTION:
Screening of people with breast tumors, through breast color Doppler ultrasound examination, the results showed that there is only a single tumor on either side of the breast. The computer tomography photoacoustic breast imaging system was used to perform breast examination again. By comparing ultrasound and photoacoustic vascular imaging, the vascular imaging of the computer tomography photoacoustic breast imaging system developed by Union Photoacoustic technologies Co., Ltd was evaluated.

This test does not evaluate the diagnosis or treatment performance of two imaging modalities. It only compares the vascular imaging of two different imaging systems. Therefore, the evaluation index of this experiment is the percentage of blood vessel pixel number in the same region of interest (ROI) to the total pixel number in ROI. By comparing the percentages of blood vessel pixel number to the total pixel number in the same ROI in ultrasound and computerized tomography photoacoustic breast imaging system, the vascular imaging of the computerized tomography photoacoustic breast imaging system is evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects aged ≥18 years old;
2. Those who have undergone breast color Doppler ultrasound examination in this hospital, and the results show that there is only a single tumor on either side of the breast;
3. Able to comply with the research procedures specified in this program;
4. Those who have fully understood the study before the experiment, volunteered to participate in the study and signed a written informed consent.

Exclusion Criteria:

1. Those with incomplete skin (such as scratches, open wounds, ulcers, etc.) in the assessment side breast area;
2. Those who have a history of surgery in the assessment side breast area;
3. Those with persistent or active breast and/or axillary infection on the assessment side;
4. Those who have a history of mental illness and cannot cooperate to complete the trial at present;
5. Subjects deemed unsuitable by the investigator to participate in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast ultrasound results suggest that there is only a single mass on either side of the breast
Sampling Method: Non-Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2021-03-31 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
ROI percentage | Immediately After photoacoustic inspection
  The evaluation index of this experiment is the percentage of blood vessel pixel number in the same region of interest (ROI) to the total pixel number in ROI

CONTACTS AND LOCATIONS:
Overall Officials: Yuxin Jiang, Doctor, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided